CLINICAL TRIAL: NCT05097625
Title: A Prospective Cohort Study of Patients With Radically Treated Newly Diagnosed Locally Advanced HPV Negative Head and Neck Cancer to Develop and Validate a Multimodal Signature to Risk-stratify for Recurrence
Brief Title: Head and Neck Early Relapse Detection Study (HERD)
Acronym: HERD
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: 277885
Record Dates: First submitted 2021-09-08; First posted 2021-10-28 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, tumour samples, saliva.
  Once used, samples will be destroyed, unless a participant has given consent for the remaining samples to be used in future similar studies, in which case these samples will be retained in a biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Risk Pathway: Risk-stratified surveillance pathway, including non-invasive methods of surveillance such as blood and saliva tests; to monitor for relapse, with any abnormalities triggering imaging
- Low Risk Pathway: Risk-stratified surveillance pathway, including non-invasive methods of surveillance such as blood and saliva tests; to monitor for relapse, with any abnormalities triggering imaging

SUMMARY:
Head and neck squamous cell carcinoma is the 6th most common cancer worldwide with an annual incidence of 12000 cases in the UK alone. More than 60% of cases are diagnosed at the locally advanced stage. These patients are treated with radical intent, using a combination of surgery, radiotherapy and/or chemotherapy. Unfortunately 5 in 10 patients relapse within 2 years, with most relapses occurring within the first year since treatment.

Unlike many other solid tumours, 80% of relapses occur locoregionally. Salvage surgery offers the best chance of long-term survival for patients with loco-regional recurrence, but this is only possible if the recurrence is amenable to resection. Salvage surgery has been estimated to improve survival outcomes in relapsed cancer by up to 73%. For salvage surgery to be feasible, relapses need to be detected early. Current surveillance strategies have little evidence base, with imaging often driven by clinical symptoms - often when the recurrence is no longer amenable to salvage surgery.

With this study, we will address the unmet clinical need to develop a risk-stratified surveillance pathway to enhance detection of early relapse of radically treated head and neck cancer. At present, tumour grade and biomarkers such as HPV status have offered important but insufficient information to guide surveillance strategies.

DETAILED DESCRIPTION:
AIMS: We hypothesise that risk of relapse relies on a dynamic interplay between the immune profile, tumour microenvironment, genetic signature and clinicopathological characteristics of the participant receiving treatment. Based on the recruitment of 200 participants within the study, we aim to generate sufficient evidence to guide a multi-analyte-based stratified imaging surveillance/follow up strategy to detect early relapse of cancer and improve survival. We will also develop a biorepository of data across a range of modalities to guide individualised treatment by precision medicine.

OBJECTIVES: The primary objective is to develop and validate a multimodal signature to risk-stratify participants with radically treated head and neck cancer into different surveillance pathways. Non-invasive methods of surveillance, such as blood and saliva tests, will be used to monitor for relapse, with any abnormalities triggering imaging. This will facilitate early detection of relapse and facilitate salvage surgery, leading to better survival outcomes.

DESIGN: This is a prospective cohort study of participants with newly diagnosed locally advanced HPV negative head and neck cancer, deemed to be intermediate or high risk (Figure 2A), referred to secondary care for radical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, locally advanced HNSCC, HPV negative considered as intermediate or high risk .
2. Offered radical treatment. (This includes surgery and any postoperative adjuvant/consolidation treatment, or radical chemo-radiation).
3. Age ≥ 18 years.
4. Adequate bone marrow function (nNeutrophils, platelets and haemoglobin grade 0 or 1 according to CTCAE).

Exclusion Criteria:

1. HPV positive disease.
2. Participants with concurrent malignancy.
3. Confirmed distant metastatic disease on most recent imaging scan.
4. Known Hepatitis B, C or HIV infection .
5. Contraindications to MRI (including but not limited to cardiac pacemaker, metallic implants, major claustrophobia).
6. Pregnant and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adults, aged 18 years and over with histologically confirmed, locally advanced HNSCC, who are HPV negative and considered of intermediate or high risk, and will be offered radical treatment. This includes surgery and any postoperative adjuvant/consolidation treatment, or radical chemo-radiation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Was a multimodal signature developed to risk-stratify participants with locally advanced radically treated head and neck cancer? | 4 years (data collection period)
  Yes or No

SECONDARY OUTCOMES:
Was a non-invasive method of surveillance successfully developed? | 4 years (data collection period)
  Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, Dr, Principal Investigator — University College, London
Locations (1):
- Guy's and St Thomas', London, United Kingdom

IPD SHARING:
Plan to Share IPD: No